CLINICAL TRIAL: NCT07200115
Title: Cervical Ripening Double Balloon Catheters Versus Osmotic Dilators For Cervical Preparation Before Dilation & Evacuation: A Randomized Controlled Trial
Brief Title: RCT of Cervical Ripening Double Ballon Catheter Prior to Dilation and Evacuation.
Acronym: CRDB RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000040146
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervical Preparation Prior to Dilation and Evacuation
Keywords: cervical preparation; osmotic dilators; cervical ripening double balloon catheter; dilation and evacuation
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cervical Ripening Double Balloon (CRDB) Catheter (Experimental)
  Interventions: Device: Cervical Ripening Double Balloon (CRDB) Catheter
- Osmotic Dilators (Active Comparator)
  Interventions: Device: Osmotic Dilators

INTERVENTIONS:
Device: Cervical Ripening Double Balloon (CRDB) Catheter — The physician will place a CRDB catheter for overnight cervical preparation. The CRDB catheter is comprised of two balloons that can be inflated with up to 80 mL of sterile water.
  Arms: Cervical Ripening Double Balloon (CRDB) Catheter
Device: Osmotic Dilators — Osmotic dilators (e.g., laminaria and Dilapan-S) are mechanical dilators that are placed in the cervix prior to gynecologic procedures and facilitate dilation through the slow absorption of moisture. The physician will place osmotic dilators in the standard fashion.
  Arms: Osmotic Dilators

SUMMARY:
The purpose of this study is to determine whether the overnight use of an FDA-cleared CRDB catheter is superior to the use of overnight osmotic dilators as is standard of care cervical preparation for patients presenting for dilation and evacuation (D&E). The CRDB catheter is an FDA cleared device for cervical dilation prior to labor induction at term. It has not been FDA cleared for cervical dilation in the second-trimester, however, will be used in a similar fashion to labor inductions at term. Our standard of care osmotic dilators (e.g., laminaria, Dilapan-S) are both FDA cleared for cervical dilation prior to labor induction at term or gynecologic procedures requiring cervical dilation.

DETAILED DESCRIPTION:
This study is a two-arm, non-blinded, randomized controlled trial of a cervical ripening double balloon (CRDB) catheter compared to osmotic dilators (e.g., laminaria and/or Dilapan-S) for overnight cervical preparation prior to dilation and evacuation (D&E). The primary outcome will be mean cervical dilation as assessed by the physician immediately prior to D&E.

Established patients will be approached by a member of the research team about study participation after they have provided informed consent for D&E. Allocation to the study group will be based on a 1:1 blocked randomization scheme. The participant will be informed of their assignment immediately prior to their cervical preparation procedure. Neither the physician nor the patient will be blinded to the assignment as this is not feasible given the differences in interventions.

1. Intervention Group: The physician will place a CRDB catheter as directed by the manufacturer's user guide. The uterine balloon of the CRDB catheter will be inflated with 20-40 mL of saline based upon the participant's tolerance.
2. Control Group: The physician will place osmotic dilators in the standard fashion. The number of dilators and use of laminaria, Dilapan-S, or a combination will be determined by physician preference.

On the day of the D&E procedure, the physician will remove the cervical dilating device and measure the patient's cervical dilation. Additional data will be collected on the following items.

* Need for and amount of mechanical dilation
* Total procedure time will be calculated in minutes based on the procedure start and stop times recorded in the patient's electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 19 weeks 0 days to 23 weeks 6 days GD.
* Planning to undergo D&E with Yale Family Planning and has undergone standard informed clinical consent counseling for the procedure and signed the clinical procedure consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the active part of the study.
* English- or Spanish-speaking individual.
* Residents of the state of Connecticut.

Exclusion Criteria:

* Spontaneous or induced fetal demise.
* Multiple pregnancy.
* Preterm prelabor rupture of membranes (PPROM).
* Intraamniotic infection.
* Active genital tract infection.
* Active vaginal bleeding.
* Placenta previa or vasa previa.
* Placenta accreta spectrum.
* History of >3 cesarean deliveries.
* BMI >45 kg/m2.
* Contraindication to osmotic cervical dilator or CRDB catheter use as determined by the physician.
* Contraindication to medication used during standard of care cervical preparation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Mean Cervical Dilation | Day 1 (cervical preparation visit) to Day 2 (D&E)
  Cervical dilation will be measured in centimeters.

SECONDARY OUTCOMES:
Need for Mechanical Dilation at the Time of Procedural Abortion | Day 2 (D&E)
  This is a binary "yes/no" outcome reported as the percentage of patients needing mechanical dilation in our experimental arm compared to the active comparator arm.
Mean Total Procedure Time | Day 2 (D&E)
  Procedure time will be measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Madden, MD, Principal Investigator — Yale University
Locations (1):
- Yale Family Planning Clinic, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atad J, Hallak M, Auslender R, Porat-Packer T, Zarfati D, Abramovici H. A randomized comparison of prostaglandin E2, oxytocin, and the double-balloon device in inducing labor. Obstet Gynecol. 1996 Feb;87(2):223-7. doi: 10.1016/0029-7844(95)00389-4. PMID 8559528
- [Background] Cook Medical. Cook Cervical Ripening Balloon with Stylet.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Liu SM, Henkel A, Meza P, Shorter JM, Cahill E, Blumenthal PD, Shaw KA. Comparing transcervical balloon with osmotic dilators for cervical preparation prior to procedural abortion: A noninferiority randomized trial. Contraception. 2024 Dec;140:110550. doi: 10.1016/j.contraception.2024.110550. Epub 2024 Jul 25. PMID 39067560
- [Background] Ornat L, Alonso-Ventura V, Bueno-Notivol J, Chedraui P, Perez-Lopez FR; Health Outcomes and Systematic Analyses (HOUSSAY) Research Group. Misoprostol combined with cervical single or double balloon catheters versus misoprostol alone for labor induction of singleton pregnancies: a meta-analysis of randomized trials. J Matern Fetal Neonatal Med. 2020 Oct;33(20):3453-3468. doi: 10.1080/14767058.2019.1574741. Epub 2019 Feb 10. PMID 30741051
- [Background] Solt I, Frank Wolf M, Ben-Haroush S, Kaminskyi S, Ophir E, Bornstein J. Foley catheter versus cervical double balloon for labor induction: a prospective randomized study. J Matern Fetal Neonatal Med. 2021 Apr;34(7):1034-1041. doi: 10.1080/14767058.2019.1623776. Epub 2019 Jun 11. PMID 31185762
- [Background] Hoppe KK, Schiff MA, Peterson SE, Gravett MG. 30 mL Single- versus 80 mL double-balloon catheter for pre-induction cervical ripening: a randomized controlled trial. J Matern Fetal Neonatal Med. 2016;29(12):1919-25. doi: 10.3109/14767058.2015.1067297. PMID 26302817
- [Background] Cook Medical. (2021) A nonpharmaceutical option for preinduction dilation. Cervical ripening balloon with stylet.
- [Background] Atad J, Hallak M, Ben-David Y, Auslender R, Abramovici H. Ripening and dilatation of the unfavourable cervix for induction of labour by a double balloon device: experience with 250 cases. Br J Obstet Gynaecol. 1997 Jan;104(1):29-32. doi: 10.1111/j.1471-0528.1997.tb10644.x. PMID 8988692
- [Background] Beaty O 3rd, Sloop CH, Schmid HE Jr, Buckalew VM Jr. Renin response and angiotensinogen control during graded hemorrhage and shock in the dog. Am J Physiol. 1976 Oct;231(4):1300-7. doi: 10.1152/ajplegacy.1976.231.4.1300. PMID 984215
- [Background] Embrey MP, Mollison BG. The unfavourable cervix and induction of labour using a cervical balloon. J Obstet Gynaecol Br Commonw. 1967 Feb;74(1):44-8. doi: 10.1111/j.1471-0528.1967.tb03931.x. No abstract available. PMID 6018096
- [Background] "Options for second-trimester termination." Contemporary OB/GYN, Nov. 2013, www.contemporaryobgyn.net/view/options-second-trimester-termination. Accessed 16 Mar. 2025.
- [Background] Lambert SJ, Lunde B, Porsch L, Stoffels G, MacIsaac L, Dayananda I, Dragoman MV. Adjuvant misoprostol or mifepristone for cervical preparation with osmotic dilators before dilation and evacuation. Contraception. 2024 Apr;132:110364. doi: 10.1016/j.contraception.2024.110364. Epub 2024 Jan 11. PMID 38218312
- [Background] White KO, Jones HE, Shorter J, Norman WV, Guilbert E, Lichtenberg ES, Paul M. Second-trimester surgical abortion practices in the United States. Contraception. 2018 Apr 14:S0010-7824(18)30140-9. doi: 10.1016/j.contraception.2018.04.004. Online ahead of print. PMID 29665357
- [Background] Casey FE, Ye PP, Perritt JD, Moreno-Ruiz NL, Reeves MF. A randomized controlled trial evaluating same-day mifepristone and misoprostol compared to misoprostol alone for cervical preparation prior to second-trimester surgical abortion. Contraception. 2016 Aug;94(2):127-33. doi: 10.1016/j.contraception.2016.02.032. Epub 2016 Mar 4. PMID 26948184
- [Background] Goldberg AB, Fortin JA, Drey EA, Dean G, Lichtenberg ES, Bednarek PH, Chen BA, Dutton C, McKetta S, Maurer R, Winikoff B, Fitzmaurice GM. Cervical Preparation Before Dilation and Evacuation Using Adjunctive Misoprostol or Mifepristone Compared With Overnight Osmotic Dilators Alone: A Randomized Controlled Trial. Obstet Gynecol. 2015 Sep;126(3):599-609. doi: 10.1097/AOG.0000000000000977. PMID 26196084
- [Background] Shaw KA, Shaw JG, Hugin M, Velasquez G, Hopkins FW, Blumenthal PD. Adjunct mifepristone for cervical preparation prior to dilation and evacuation: a randomized trial. Contraception. 2015 Apr;91(4):313-9. doi: 10.1016/j.contraception.2014.11.014. Epub 2014 Dec 12. PMID 25499589
- [Background] Diedrich JT, Drey EA, Newmann SJ. Society of Family Planning clinical recommendations: Cervical preparation for dilation and evacuation at 20-24 weeks' gestation. Contraception. 2020 May;101(5):286-292. doi: 10.1016/j.contraception.2020.01.002. Epub 2020 Jan 31. PMID 32007418
- [Background] Sanchez-Ramos L, Levine LD, Sciscione AC, Mozurkewich EL, Ramsey PS, Adair CD, Kaunitz AM, McKinney JA. Methods for the induction of labor: efficacy and safety. Am J Obstet Gynecol. 2024 Mar;230(3S):S669-S695. doi: 10.1016/j.ajog.2023.02.009. Epub 2023 Jul 13. PMID 38462252